CLINICAL TRIAL: NCT03450746
Title: Metabolic and Physiological Changes During Minor Orthopaedic Surgery in Otherwise Healthy Patients
Status: Completed | Type: Observational
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Bodil Steen Rasmussen, Professor, Aalborg University Hospital
Other Study IDs: AAUH-ANAESTH-03
Record Dates: First submitted 2017-12-22; First posted 2018-03-01 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Metabolomics; Anesthesia, General; Oxygen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Exhaled breath condensate and arterial blood for matabolomic analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy patients for orthopaedic surgery: Standard general anaesthesia and ventilation with FiO2 0.50 for at least 45 minutes following the standard settings in our department.

SUMMARY:
The air we breathe contains 21% of oxygen. Oxygen is vital for the cells ability to produce energy and without it we could not survive. Oxygen normally exists as a molecule consisting of two atoms, O2. It has two unpaired electrons and thus is unstable and willing to accept electrons to become stable. During the formation of ATP a transportation of electrons happens over the inner membrane of the mitochondria's. Oxygen can accept these and is thereby reduced to water. Normally about 4% is not fully reduced and instead produces superoxide. Superoxide is transformed to hydrogen peroxide by superoxide dismutase (SOD) and then into oxygen and water by catalase and glutathione peroxidase. It is also possible for hydrogen peroxide to be converted to hydroxyl radicals by Fenton reactions. All these radicals are called reactive oxygen species (ROS) and they are highly reactive and capable to induce damage to cellular components as proteins, DNA and lipids. Under normal conditions SOD, catalase and glutathione peroxidase work as anti-oxidative compounds to prevent oxidative stress and damage. However, under hyperoxic conditions these defences can be overwhelmed, resulting in the formation of excess ROS and thus oxidative damage.

During general anaesthesia the use of supplemental oxygen to avoid life-threatening hypoxaemia has been common practice for many years and a fixed fraction of inspired oxygen (FiO2) ranging from 0.3 to 1.0 is often used. This lead to supranormal levels of oxygen in the lungs and most of the patients also have supranormal levels of partial pressure of arterial oxygen in their blood.

This study will examine otherwise healthy ambulant patients undergoing minor orthopaedic surgery during general anaesthesia to elucidate metabolic and physiological changes caused by ventilation with FiO2 0.50 for at least 45 minutes using standard respiratory settings. Exhaled breath condensate (EBC) and arterial blood will be collected prior to and after surgery. The two EBCs and two blood samples will be stored at -80°C for analysis after all patients have been included. The metabolic changes will be measured with NMR technique and multivariate statistical analysis comparing baseline values with values obtained after oxygen exposure.

Collapse of the small airways induced by anaesthesia and FiO2 will be evaluated by measuring resistance and reactance with airway oscillometry after surgery compared to a baseline measurement before surgery.

DETAILED DESCRIPTION:
Oxygen supplement during general anaesthesia During general anaesthesia the use of supplemental oxygen to avoid life-threatening hypoxaemia has been common practice for many years. This lead to supranormal levels of oxygen in the lungs (hyperoxia) and most patients also have supranormal levels of partial pressure of arterial oxygen (PaO2) in their blood (hyperoxaemia). The same iatrogen hyperoxia is also common in mechanically ventilated patients in the intensive care unit. Is seems to be forgotten that supplemental oxygen is a medicine and like all medication it should not be administered in excess.

During general anaesthesia a fixed fraction of inspired oxygen ranging from 0.3 to 1.0 is often used. Patients are monitored with continuously measurement of peripheral oxygen saturation and if this is low or an arterial gas shows low PaO2 then FiO2 is further increased. However, a decrease beyond the prefixed FiO2 is seldom done even if oxygen saturation is 100% or the arterial gas shows a high PaO2.

More and more evidence question the safety of this liberal use of hyperoxia as high oxygen supplement and the formation of ROS can lead to cell dysfunction and thereby contribute to pulmonary dysfunction postoperatively.

Adverse effects of oxygen FiO2 exceeding the atmospheric content of 0.21 can have direct toxic effects on lung tissue especially for FiO2 exceeding 0.60. Studies from the 1970's showed that when breathing FiO2 1.0 for more than four hours people experienced mild symptoms like tracheobronchitis and pleuritic. This is a mild irritation behind the sternum, in the airways or in the lungs. This discomfort is aggravated by deep inspiration and can cause cough. They also showed that a high FiO2 of 0.95-1.0 given for several days lead to pulmonary edema and eventually lung fibrosis. High FiO2 also induce collapse of lung areas leading to pulmonary shunt because of reabsorption atelectasis and induce pulmonary vasodilatation but otherwise induce vasoconstriction in all others vascular beds (except in uterus) and thereby reduce cardiac output and end organ perfusion.

The precise mechanism of the direct cellular damage and vasoconstriction is unknown but is believed to be due to increased production of ROS5.

In the clinical setting with critical ill patients hyperoxia and hyperoxaemia has been associated with increased mortality specifically in subgroups of patients with stroke, traumatic brain injury and those resuscitated from cardiac arrest and it is also shown to increased infarct size and mortality after cerebral and myocardial infarction. Perioperative treatment with high FiO2 has also been associated with increased mortality and major respiratory complications.

Metabonomics Lately there has been a lot of attention on the formation of ROS during hyperoxic conditions. Besides induction oxidative stress ROS also affects a number of signal-transduction-pathways that leads to cellular changes. These changes can be detected using metabonomics.

Metabonomics is the analysis of all small molecules or metabolites present in a given sample using nuclear magnetic resonance (NMR) or mass spectrometry (MS). Metabonomics gives a "snapshot" of all metabolites in a given sample and thus has great potential to find several new biomarkers by analysis of the continuous changes in the metabolic profile in response to a given exposure.

Oscillometry Anaesthesia and high FiO2 lead to collapse of the small airways. A new airway oscillometry system (TremoFlo C-100) enables a simple and non-invasive measurement of changes in the small airways. The system measure resistance and reactance non-invasively during normal breathing.

The trial We will examine otherwise healthy ambulant patients undergoing minor orthopaedic surgery during general anaesthesia to elucidate metabolic and physiological changes caused by ventilation with FiO2 0.50 for 45 minutes following standard settings. Exhaled breath condensate (EBC) and arterial blood will be collected prior to the surgery and repeated during surgery after 45 minutes of mechanical ventilation with a FiO2 0.50. The two EBCs and two blood samples will be stored at -80°C for analysis after all patients have been included. The metabolic changes will be measured with NMR technique and multivariate statistical analysis comparing baseline values with values obtained after 45 minutes of oxygen exposure. All specimens will be destroyed after the NMR analyses. Collapse of the small airways induced by anaesthesia and FiO2 will be evaluated by measuring resistance and reactance after surgery compared to a baseline measurement before surgery.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 18 years
* Otherwise healthy (No major illness and not taking any medicine on a regular basis)
* Non-smoker (Have never smoked or stopped smoking two years or more before the trial date)
* Have given informed consent

Exclusion Criteria:

* Any respiratory infection in the past three months leading to consulting a doctor (Any infection in the lungs or the airways in the three months leading up to the trial that resulted in the participant consulting a doctor or taking any medication for the infection)
* Any alcohol intake the last 24 hours (Drinking any alcohol in the last 24 hours up to the start of the trial)
* Pregnancy (Confirmed by positive urine human gonadotropin (hCG) or plasma-hCG)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects are recruited at Aalborg University Hospital in Denmark among patients scheduled for ambulant minor orthopedic surgery expected to last at least 45 minutes.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2017-11-02 (Actual); Primary Completion 2017-11-22 (Actual); Study Completion 2017-11-22 (Actual)

PRIMARY OUTCOMES:
Metabolites in exhaled breath condensate and in arterial blood | minor surgery (approximately 45-120 minutes)
  Metabolites measured by Nuclear Magnetic Resonance spectroscopy (NMR), explanatory study thus every changes in metabolites will be visualized

SECONDARY OUTCOMES:
Minor airway resistance | minor surgery (approximately 45-120 minutes)
  Measured by oscillometry
Airway reactance | minor surgery (approximately 45-120 minutes)
  Measured by oscillometry
Mean arterial bloodpressure | minor surgery (approximately 45-120 minutes)
  Measured invasively
heart rate | minor surgery (approximately 45-120 minutes)
  changes in the heart rate meassured 30 minutes after the awakening from general anaesthesia compaired to baseline (30 minutes before surgery)
oxygen saturation | minor surgery (approximately 45-120 minutes)
  changes in the oxygen saturation meassured 30 minutes after the awakening from general anaesthesia compaired to baseline (30 minutes before surgery)
Partial pressure of arterial oxygen | minor surgery (approximately 45-120 minutes)
  Measured with blodgas analyzer (Radiometer, Denmark)

CONTACTS AND LOCATIONS:
Overall Officials: Bodil S Rasmussen, Professor, Principal Investigator — Department of Anaesthesia and Intensive Care Medicine, Aalborg University Hospital
Locations (1):
- Departmen of Anaesthesia and Intensive Care Medicine, Aalborg University Hospital, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No